CLINICAL TRIAL: NCT00604266
Title: Coregistration of 18F-FDG-PET and MRI in the Staging of Potentially Resectable Hilar Cholangiocarcinoma: a Pilot Study.
Acronym: PET/MRCP
Status: Withdrawn | Type: Observational
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ur Metser, Division Head, Molecular Imaging, Joint Department of Medical Imaging, University of Toronto
Other Study IDs: 07-0216
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Cholangiocarcinoma
Keywords: Potentially resectable hilar cholangiocarcinoma as per initial imaging studies.; Able to undergo PET/CT and MRI with Gadolinium
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: 10-15 patients with potentially resectable hiilar cholangiocarcinoma

SUMMARY:
To evaluate the feasibility and performance of coregistered 18F-FDG-PET/MRI in the staging of potentially respectable hilar cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Hilar cholangiocarcinoma assessed by conventional imaging modalities (triphasic CT scan of the liver) and thought to be potentially resectable.

Exclusion Criteria:

* Biliary drain inserted.
* Contraindication for MRI.
* Pregnant or breast-feeding.
* Uncontrolled diabetes (over 9.7 mmol/L).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifteen patients with potentially resectable hilar cholangiocarcinomas, as determined by conventional imaging modalities, will be recruited. In order to minimize false positive uptake of 18F-FDG due to inflammatory changes, patients will be recruited either before biliary stenting, or after biliary stenting if there is no clinical evidence of active cholangitis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ur Metser, MD, Principal Investigator — U of Toronto, UHN
Locations (1):
- UHN - Princess Margaret Hospital, Toronto, Ontario, Canada